CLINICAL TRIAL: NCT04360031
Title: Investigating the Links Between Microbiota Composition and Variability Observed in the Pharmacological Response to Immunosuppressive Therapies in Kidney Transplant Patients.
Brief Title: The Effects of Microbiota Composition on Immunosuppression Protocols in Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: Microbiota/TAC/MPA
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-02

CONDITIONS: Kidney Transplant; Complications; Immunosuppression; Transplant Failure
Keywords: Tacrolimus; Mycophenolate Mofetil; Transplantation; Kidney transplant; Calcineurin inhibitors
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In all patients, blood and urine will be retained, Feces samples will be collected and retained(when possible),
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: No

GROUPS / COHORTS (1):
- Tacrolimus / Mycophenolate Mofetil: All patients receive maintenance immunosuppressive treatment of tacrolimus in combination with Mycophenolate Mofetil.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus and Mycophenolate Mofetil are given in accordance with patient's current regimen
  Other Names: Mycophenolate Mofetil

SUMMARY:
Solid organ transplantation is the treatment of choice for patients suffering from end-stage organ disease, including for chronic kidney failure. The implementation of effective immunosuppressive therapies has already significantly improved the prognosis for graft survival. However, these therapies are often associated with considerable inter- and intra-individual variability both in terms of response or in terms of pharmacokinetics. Innovative approaches must be considered, such as studying the involvement of intestinal microbiota in the pharmacology of these drugs.

The general aim of the study is therefore to relate the variabilities observed in the pharmacology (mainly pharmacokinetics) of immunosuppressive drugs used in renal transplantation (tacrolimus and mycophenolate mofetil) and the composition of the intestinal microbiota of renal transplant patients.

DETAILED DESCRIPTION:
Solid-organ transplantation often requires the implementation of a lifelong immunosuppressive therapy. A combination of tacrolimus (TAC), mycophenolate mofetil (MMF), together with steroids is currently used in over 60% of cases. In some patients however, these therapies are associated with high levels of variability, either in terms of response to treatments or in terms of pharmacokinetics, which remains unexplained. To address the issue, new approaches are being considered, in this study we will investigate the involvement of the intestinal microbiota in the pharmacology of these drugs. This is a particularly promising avenue for drugs with a low therapeutic index and large intra- and inter-individual pharmacokinetic variabilities such as tacrolimus and mycophenolate mofetil. Despite promising preliminary data for tacrolimus, the influence of the gut microbiota in these pharmacokinetic variabilities remains unclear, even less data are available about the involvement of the microbiota in the pharmacokinetics of mycophenolate mofetil.

We expect that this study will produce additional information on the effect of immunosuppression drugs on gut microbiota, and the relationship between microbiota composition and variabilities.

ELIGIBILITY:
Inclusion Criteria:

* Patients within 1 to 8 years post transplantation
* Aged between 18 and 75 years old
* Patients receiving tacrolimus and mycophenolate mofetil as part of their immunosuppressive therapy
* French speaking
* BMI between 18 and 30.

Exclusion Criteria:

* Use of tobacco
* Potential Alcohol problems (less than two positive answers to the CAGE questionnaire)
* Use of antibiotic medication within 3 months of the sample collection
* Use of laxative medication within 2 weeks of the sample collection
* Use of anti-fungal medication within 2 weeks of the sample collection
* Pregnant or lactating patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant patients followed at the Saint-Luc University Clinics and having been transplanted in the abdominal transplant service of the clinics will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Study of the links between immunosuppressive drugs pharmacology and intestinal microbiota composition | 24 months
  The general aim of the study is to relate the variabilities observed in the pharmacology (mainly pharmacokinetics) of immunosuppressive drugs used in kidney transplantation (tacrolimus and mycophenolate mofetil) and the composition of the intestinal microbiota of these patients.

SECONDARY OUTCOMES:
Identify links between oral dosage and concentrations found in feces | 18 months
  Study the concentrations of Tacrolimus and Mycophenolate (MPA) Mofetil in feces and highlight predictors depending on microbiota composition
Identify genetic factors underlying the links between microbiota and Tacrolimus/Mycophenolate Mofetil | 18 months
  Investigate microbial genes responsible for associations between microbiota composition and immuno-suppressant pharmacology
Tacrolimus concentrations and microbiota | 18 months
  Identify links between microbiota composition and Tacrolimus concentrations in blood.
Tacrolimus concentrations and genetic polymorphisms | 18 months
  Identify genetic factors able to influence Tac concentrations in blood.
Tacrolimus concentration and demographics | 18 months
  Investigate the effect of sex and age on Tac concentrations in blood.
Mycophenolate Mofetil concentration and microbiota | 18 months
  Identify links between microbiota composition and MPA Mofetil concentration in blood and urine.
Mycophenolate Mofetil concentration and polymorphisms | 18 months
  Identify genetic factors able to influence MPA Mofetil concentrations in blood and urine.
Mycophenolate Mofetil concentration and demographics | 18 months
  Investigate the effect of sex and age on MPA Mofetil concentrations in blood and urine.
Investigate potential markers of kidney function in metabolites | 18 months
  Study metabolomics in urine from patients to identify specific markers of kidney function

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Haufroid, MD, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Degraeve AL, Bindels LB, Haufroid V, Moudio S, Boland L, Delongie KA, Dewulf JP, Eddour DC, Mourad M, Elens L. Tacrolimus Pharmacokinetics is Associated with Gut Microbiota Diversity in Kidney Transplant Patients: Results from a Pilot Cross-Sectional Study. Clin Pharmacol Ther. 2024 Jan;115(1):104-115. doi: 10.1002/cpt.3077. Epub 2023 Oct 30. PMID 37846607